CLINICAL TRIAL: NCT07206745
Title: Efficacy Evaluation of Integrated Traditional Chinese and Western Medicine in the Treatment of Severe Pneumonia Caused by Multidrug-Resistant Gram-Negative Bacterial Infections: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Study on Integrated Chinese and Western Medicine for Severe Pneumonia Caused by Multidrug-Resistant Gram-Negative Bacterial Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Henan Provincial Hospital of TCM (Unknown); Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for MDR-GNB pneumonia
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Severe Pneumonia Caused by Multidrug-resistant Gram-negative Bacterial Infection
Keywords: Severe pneumonia; multidrug-resistant Gram-negative bacterial infection; traditional Chinese medicine; randomized controlled trial; Fei Re Qing Granules
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The patients in the trial group received routine standard treatments, and oral Fei Re Qing Granules (One bag/time, 3 times/day).
  Interventions: Drug: Fei Re Qing Granules
- Control group (Placebo Comparator): The patients in the control group received routine standard treatments, and Placebo granules
  Interventions: Drug: Placebo of Feireqing Granules

INTERVENTIONS:
Drug: Fei Re Qing Granules — Fei Re Qing Granules (Ingredients: Scutellaria baicalensis [Huang Qin], Trichosanthes kirilowii [Gua Lou], Forsythia suspensa [Lian Qiao], Fritillaria thunbergii [Zhe Bei Mu], etc.).
  Routine standard treatments：Routine standard treatments according to clinical guidelines.
  Arms: Test group
Drug: Placebo of Feireqing Granules — Placebo of Feireqing Granules：The placebo granules are prepared using 5% of the active drug combined with pharmaceutical excipients, including starch, dextrin, microcrystalline cellulose, and food-grade coloring and flavoring agents, to ensure consistency in appearance, weight, color, and odor with the Fei Re Qing Granules.
  Routine standard treatments：Routine standard treatments according to clinical guidelines.
  Arms: Control group

SUMMARY:
This study aims to evaluate the clinical efficacy of a traditional Chinese medicine formula granule (Feireqing Granules) in the treatment of severe pneumonia caused by multidrug-resistant Gram-negative bacterial infections (MDR-GNB severe pneumonia), to establish a therapeutic regimen, and to generate high-quality clinical evidence.

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of Feireqing Granules for MDR-GNB severe pneumonia through a multicenter, randomized, double-blind, placebo-controlled trial.

Key elements of the trial include:

Design: Conducted across multiple centers, comparing Feireqing Granules and placebo groups, alongside standard guideline-based modern medical treatment.

Participants: Patients diagnosed with MDR-GNB severe pneumonia according to modern medical diagnostic criteria, aged ≥18 years and <80 years. 76 patients will be enrolled in each group.

Intervention:

Test group: Participants will receive Feireqing Granules in combination with standard modern medical treatments.

Control group: Participants will receive placebo granules (matching the appearance, weight, color, and odor of the active granules, composed mainly of starch, dextrin, microcrystalline cellulose, and 5% active drug) in combination with standard modern medical treatments.

Outcomes:

Primary efficacy indicator: All-cause mortality.

Secondary indicators: Clinical cure rate, bacterial clearance rate, duration of antibiotic therapy, effective mechanical ventilation rate, length of hospital stay, Clinical Pulmonary Infection Score (CPIS), Acute Physiology and Chronic Health Evaluation II (APACHE II) score, and Sequential Organ Failure Assessment (SOFA) score.

Study Duration: Treatment for 14 days, with a 28-day follow-up.

This trial seeks to confirm the clinical efficacy of Feireqing Granules in treating MDR-GNB severe pneumonia and to provide high-quality evidence for the long-term and objective evaluation of TCM interventions.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for severe pneumonia, aged ≥18 years and <80 years;
* Microbiological culture confirming Gram-negative bacterial infection resistant to three or more classes of antibiotics, such as extended-spectrum β-lactamase (ESBL)-producing Enterobacteriaceae, carbapenem-resistant Enterobacteriaceae, carbapenem-resistant Acinetobacter baumannii (CRAB), and multidrug-resistant Pseudomonas aeruginosa (MDR-PA);
* Written informed consent obtained from the patient or their legal representative.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Patients with impaired consciousness, dementia, psychiatric disorders, or other conditions that preclude effective communication and cooperation;
* Patients with aspiration pneumonia, fungal pneumonia, viral pneumonia, pulmonary tuberculosis, or HIV-associated Pneumocystis jirovecii pneumonia;
* Patients with severe hepatic or renal insufficiency, such as liver cirrhosis with Child-Pugh score of 10-15, or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²;
* Patients with hematologic malignancies, solid organ transplantation, or congenital/acquired diseases leading to immunodeficiency;
* Patients with multidrug-resistant bacterial infections outside the lung (e.g., urinary tract, abdominal cavity, bloodstream);
* Patients with severe cardiac dysfunction (NYHA class IV), malignant arrhythmias, or other hemodynamically unstable conditions;
* Patients who have already received antimicrobial therapy for more than one week;
* Patients who have participated in another drug clinical trial within one month prior to enrollment;
* Patients with known allergy to the investigational drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | All-cause mortality: assessed at 14 and 28 days post-enrollment.
  All-cause mortality will be assessed as the proportion of participants who die from any cause during the study period. Mortality will be recorded at Day 14 and Day 28 after enrollment.

SECONDARY OUTCOMES:
Clinical cure rate | Evaluations will be conducted on treatment Day 0, Day 14 and during follow-up on Day 28.
  According to the Technical Guidelines for Clinical Trials of Antibacterial Drugs, clinical cure is defined as the complete resolution or normalization of all symptoms and signs present at baseline at the post-treatment visit, along with normalization of non-microbiological indicators such as imaging and laboratory tests. In practice, some clinical symptoms or signs, or abnormalities in non-microbiological indicators, may still be observed at the post-treatment visit. If these findings are physiological, reflect post-infection status, or are related to underlying diseases rather than active infection, they may also be considered indicative of clinical cure.
Bacterial clearance rate | Treatment days 0, days 7, and days 14.
  Based on microbiological testing during hospitalization. Pathogen-targeted next-generation sequencing (tNGS) of bronchoalveolar lavage fluid or sputum, or sputum culture, is performed on treatment days 0, 7, and 14 for evaluation.
Duration of antibiotic use | From Day 0 of treatment to Day 28 of follow-up
  Total number of days of antibiotic therapy during hospitalization, including both intravenous and oral administration.
Invasive mechanical ventilation rate | From Day 0 of treatment to Day 28 of follow-up
  The invasive mechanical ventilation rate will be assessed as the proportion of participants who require invasive mechanical ventilation during the study period. Eligible participants are those not receiving invasive ventilation at baseline (Day 0). The outcome is defined as the need for endotracheal intubation and mechanical ventilation due to clinical deterioration, including worsening hypoxemia, hypercapnia, or respiratory failure. The rate will be calculated as the number of participants requiring invasive mechanical ventilation divided by the total number of participants at risk, from Day 0 of treatment to Day 28 of follow-up.
Length of hospital stay | From Day 0 of treatment to Day 28 of follow-up
  Total number of days of hospitalization
Clinical Pulmonary Infection Score (CPIS) | Assessed on treatment days 0, 7, and 14, and on follow-up days 14 and 28.
  The Clinical Pulmonary Infection Score (CPIS) will be used to evaluate the presence and severity of pulmonary infection. The CPIS is calculated based on a composite of clinical, radiological, and laboratory parameters, including body temperature, leukocyte count, tracheal secretions, oxygenation (PaO₂/FiO₂), chest radiograph findings, and culture results of tracheal aspirate. Each component is scored from 0 to 2 points, with a maximum total score of 12; higher scores indicate more severe infection. CPIS will be assessed on treatment days 0, 7, and 14, as well as on follow-up days 14 and 28.
SOFA score | Recorded on treatment days 0, 7, and 14, and on follow-up days 14 and 28.
  The Sequential Organ Failure Assessment (SOFA) score will be used to evaluate the extent of organ dysfunction during the study. The SOFA score includes six components: respiratory function (PaO₂/FiO₂ ratio), coagulation (platelet count), liver function (bilirubin), cardiovascular status (mean arterial pressure or vasopressor requirement), central nervous system function (Glasgow Coma Scale), and renal function (serum creatinine or urine output). Each organ system is scored from 0 (normal) to 4 (severe dysfunction), with a total score ranging from 0 to 24. Higher scores indicate more severe organ dysfunction and higher risk of mortality. SOFA scores will be assessed on treatment days 0, 7, and 14, and on follow-up days 14 and 28.
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | From Day 0 of treatment to Day 28 of follow-up
  The Acute Physiology and Chronic Health Evaluation II (APACHE II) score will be used to evaluate the severity of illness and the risk of mortality. The score incorporates the acute physiology score, age score, and chronic health score. Higher total scores indicate more severe illness and greater mortality risk. APACHE II scores will be recorded on treatment days 0, 7, and 14, and on follow-up days 14 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine